CLINICAL TRIAL: NCT06706102
Title: Temporal Characterization of Extracellular Vesicles During Cellular Therapy Using CAR-T Cells and During the Occurrence of Immune Effector Cell-Associated Neurotoxicity Syndrome
Acronym: VESICANS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24CH009; 2024-515328-35-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-14; First posted 2024-11-26 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Immune Effector Cell Associated Neurotoxicity Syndrome
Keywords: CAR-T Cell; ICANS; EVs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR T cell treatment (Experimental): Major patients for whom CAR-T treatment is indicated.
  Interventions: Biological: Biological tests; Diagnostic Test: MRI; Diagnostic Test: Neuropsychological tests

INTERVENTIONS:
Biological: Biological tests — Biological tests : cell quantification et characterization
Diagnostic Test: MRI — MRI
Diagnostic Test: Neuropsychological tests — Neuropsychological tests

SUMMARY:
Immune effector Cell-Associated Neurotoxicity Syndrome (ICANS) is a common and serious neurological complication associated with the use of CAR-T cells. The mechanisms involved are still poorly understood but studies suggest that inflammation during treatment leads to an increase in the permeability of the barrier between the brain and the blood vessels and the emission of extracellular vesicles (EVs) circulating between the brain and the blood vessels. EVs are biological particles that play an important role in cellular communication and the modulation of several physiological processes. The VESICANS study aims to characterize the EVs released before and during CAR-T cells treatment and upon the occurrence of ICANS, using flow cytometry, electron microscopy, Nanoparticle Tracking Analysis associated with MRI assessment of the barrier between the brain and blood. This study will ultimately contribute to facilitating the prevention and treatment of this toxicity which affects the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18,
* Patient for whom CAR-T treatment is indicated,
* Patient affiliated to a social security system
* Patient who give his consent to participate in the study.

Exclusion Criteria:

* Pregnant or breastfeeding woman,
* Patient unable to understand informed consent,
* Patient under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Endothelial EVs quantification (EVs/mL) | Days -7, 0, 1, 2, 5, 8, 15, 30 and 60
  Quantification by Nano Tracking Analysis of endothelial EVs as a function of time before and after treatment with CAR-T cells according to ICANS grade.
Endothelial EVs characterization (immunophenotyping) | Days -7, 0, 1, 2, 5, 8, 15, 30 and 60
  Characterization by Nano Tracking Analysis (immunophenotyping by size) of endothelial EVs as a function of time before and after treatment with CAR-T cells according to ICANS grade.

SECONDARY OUTCOMES:
Other EV subtypes quantification (EV subtype/mL) | Days -7, 0, 1, 2, 5, 8, 15, 30 and 60
  Other EV subtypes quantification of as a function of time before and after treatment with CAR-T cells according to ICANS grade.
Other EV subtypes characterization (immunophenotyping) | Days -7, 0, 1, 2, 5, 8, 15, 30 and 60
  Other EV subtypes characterization of as a function of time before and after treatment with CAR-T cells according to ICANS grade.
EVS quantification according to the presence of an ICANS versus no ICANS (EV/mL) | Days -7, 0, 1, 2, 5, 8, 15, 30 and 60
  EVS quantification according to the presence of an ICANS versus no ICANS
EVs characterization according to the presence of an ICANS versus no ICANS (immunophenotyping) | Days -7, 0, 1, 2, 5, 8, 15, 30 and 60
  EVS characterization of EVs according to the presence of an ICANS versus no ICANS
EVs quantification according to levels of cytokines (EVs/mL) | Days -7, 0, 1, 2, 5, 8, 15, 30 and 60
  EVs quantification according to levels of cytokines
EVs characterization according to levels of cytokines | Days -7, 0, 1, 2, 5, 8, 15, 30 and 60
  EVs characterization according to levels of cytokines
EVs quantification in cerebrospinal fluid (EVs/mL) | Days -7, 0, 1, 2, 5, 8, 15, 30 and 60
  EVs quantification after treatment with CAR-T cells in cerebrospinal fluid (CSF) if available.
EVs characterization in cerebrosinalfluid. | Days -7, 0, 1, 2, 5, 8, 15, 30 and 60
  EVs characterization of EVs after treatment with CAR-T cells in cerebrospinal fluid (CSF) if available.
Association of EVs subpopulations in clinical neurological damage and sleep apnea syndrome. | Days -7, 0, 1, 2, 5, 8, 15, 30 and 60
  Characterization of the association of subpopulations of EVs according to clinical neurological damage and sleep apnea syndrome.
Association of EVs subpopulations in neuropsychological test and RMI. | Days -7, 0, 1, 2, 5, 8, 15, 30 and 60
  Characterization of the association of subpopulations of EVs according to neuropsychological test and RMI.
Cerabral involvement on RMI | Days -7, 0, 1, 2, 5, 8, 15, 30 and 60
  Diffusion tensor imaging and resting state default mode network

CONTACTS AND LOCATIONS:
Overall Officials: Emilie CHALAYER, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No